CLINICAL TRIAL: NCT00154206
Title: A Multicenter, Open, Single Arm, Pilot Study to Evaluate Efficacy, Tolerability and Safety of Enteric-Coated Mycophenolate Sodium (EC-MPS) in Combination With Cyclosporine Microemulsion and Steroids in Pediatric de Novo Renal Transplant Patients
Brief Title: Study of Enteric-coated Mycophenolate Sodium (EC-MPS) With Cyclosporine Microemulsion and Steroids in Pediatric de Novo Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080AFR03
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplantation
Keywords: Enteric-coated mycophenolate sodium,; de novo,; renal transplantation,; pediatric; De novo pediatric renal transplantation

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
The aim of this pilot study is to evaluate efficacy and tolerability of EC-MPS b.i.d, with Cyclosporine microemulsion and steroids in pediatric de novo renal transplant patients. Safety and doses variations are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a primary renal transplantation
* Recipients of a renal transplantation only

Exclusion Criteria:

* Recipients of a multi-organ transplantation
* Unable to take an oral medication
* Requiring an induction therapy with polyclonal, monoclonal antibodies (OKT3, ATG, ALG).

Other protocol-defined inclusion / exclusion criteria may apply

Ages: 5 Years to 16 Years | Sex: All
Age Groups: Child
Enrollment: 15
Dates: Start 2004-09; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy-proven-acute-rejection and treatment failure (defined by graft loss and/or biopsy-proven-acute-rejection and/or death and/or lost to follow-up and/or study discontinuation) within the 6 and 12 months post transplantation

SECONDARY OUTCOMES:
Within the 6 and 12 months post transplantation
Incidence of acute rejection resistant to steroids
Incidence of graft loss and death
Renal function by creatinine and creatinine clearance (Schwartz formula)
Incidence of premature study drug discontinuation due to safety reason
Pharmacokinetic profile of Myfortic.
Frequency of adverse events, incidence of clinically notable laboratory abnormalities, and change on vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Background] Niaudet P, Charbit M, Loirat C, Lapeyraque AL, Tsimaratos M, Cailliez M, Foulard M, Dehennault M, Marquet P, Chaouche-Teyara K, Lemay D. Enteric-coated mycophenolate sodium in de novo pediatric renal transplant patients. Pediatr Nephrol. 2009 Feb;24(2):395-402. doi: 10.1007/s00467-008-1031-7. Epub 2008 Nov 5. PMID 18985393